CLINICAL TRIAL: NCT05025332
Title: An Open-Label Study of the Safety, Tolerability, and Pharmacokinetics of Oral NNZ-2591 in Pitt Hopkins Syndrome (PTHS-001)
Brief Title: An Open-Label Study of Oral NNZ-2591 in Pitt Hopkins Syndrome (PTHS-001)
Acronym: PTHS-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-2591-PTHS-001
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pitt Hopkins Syndrome
Keywords: Pitt Hopkins Syndrome
MeSH Terms: conditions — Pitt-Hopkins syndrome | interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNZ-2591 (Experimental): NNZ-2591 oral solution (50mg/mL) to be administered twice daily dose for 13 weeks.
  Interventions: Drug: NNZ-2591

INTERVENTIONS:
Drug: NNZ-2591 — NNZ-2591 oral solution (50mg/mL) to be administered twice daily dose for 13 weeks.
  Other Names: Cyclo-L-Glycyl-L-2-Allylproline

SUMMARY:
A study of the safety, tolerability and pharmacokinetics of NNZ-2591 and measures of efficacy in children and adolescents with Pitt Hopkins Syndrome.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate the safety, tolerability and pharmacokinetics of treatment with NNZ-2591 oral solution in children and adolescents with Pitt Hopkins Syndrome. The secondary purpose is to investigate measures of efficacy. Subjects will receive treatment with NNZ-2591 oral solution (50 mg/mL) doses for a total of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PTHS with a documented disease-causing genetic etiology for the disorder.
2. Males or females aged 3-17 years.
3. Body weight of 12kg or higher at screening
4. Subjects with a Clinical Global Impression- Severity (CGI-S) score of 4 or greater at the Screening visit.
5. Not actively undergoing regression or loss of skills, defined as no persistent loss of previously acquired developmental skills for a period within 3 months of the Screening visit
6. Each subject must be able to swallow the study medication provided as a liquid solution.
7. Caregiver(s) must have sufficient English language skills.

Exclusion Criteria:

1. Body weight <12kg at screening
2. Clinically significant abnormalities in safety laboratory tests and vital signs at Screening.
3. Abnormal QTcF interval or prolongation at Screening.
4. Any other clinically significant finding on ECG at the Screening visit.
5. Positive for severe acute respiratory syndrome coronavirus 2 (SARSCoV-2) and previous COVID 19 infection with last 12 months that required hospitalization.
6. Unstable or changes Psychotropic treatment 2 weeks prior to screening
7. Excluded concomitant treatments.
8. Actively undergoing regression or loss of skills.
9. Unstable seizure profile.
10. Current clinically significant renal conditions and abnormalities
11. Current clinically significant cardiovascular, hepatic, gastrointestinal, respiratory, endocrine disease, or clinically significant organ impairment.
12. Current clinically significant hypo- or hyperthyroidism, Type 1 or Type 2 diabetes mellitus requiring insulin (whether well controlled or uncontrolled), or uncontrolled Type 1 or Type 2 diabetes.
13. Has planned surgery during the study.
14. History of, or current, cerebrovascular disease or brain trauma.
15. History of, or current catatonia or catatonia-like symptoms.
16. History of, or current, malignancy.
17. Current major or persistent depressive disorder (including bipolar depression).
18. Significant, uncorrected visual or uncorrected hearing impairment.
19. Allergy to strawberry.
20. Positive pregnancy test
21. Subject is judged by the Investigator or Medical Monitor to be inappropriate for the study

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Shaw, Study Director — Neuren Pharmaceuticals
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - UT Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 5 academic medical centers between August 2022 and December 2023
Pre-assignment Details: Following completion of informed consent, participants (28) underwent 4 weeks of baselining/screening. During this process 12 participants failed screening. The remaining 16 participants commenced treatment.
Groups:
- NNZ-2591: All participants consenting
Period: Screening
Arm/Group | NNZ-2591
Started | 28
Completed | 16
Not Completed | 12
Not completed — Screen failure | 12
Period: Treatment & Follow Up
Arm/Group | NNZ-2591
Started | 16
Completed | 11
Not Completed | 5
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Groups:
- NNZ-2591: All participants who successfully completed 4 week post consent screening period.
Arm/Group | NNZ-2591
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (4.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Black or African American | 1
  Native Hawaiian or other Pacific Islander | 0
  White | 11
  Other | 1
  Multiple | 0
  Unknown | 0
Clinical Global Impression of Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] | 5.0 (0.69)
Height (cm) [Mean (Standard Deviation); unit: centimetres] | 127.26 (22.609)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 28.57 (12.291)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 16.846 (2.0979)
PTHS variant [Number; unit: participants]
  Substitution | 5
  Deletion | 6
  Duplication | 0
  Insertion | 0
  Inversion | 0
  Conversion | 0
  Deletion-Insertion | 0
  Complex | 0
  Missense variant | 2
  Nonsense variant | 3
  Frameshift variant | 2
  Unknown | 1
  Other | 2
History of Developmental Regression [Count of Participants; unit: Participants]
  Yes | 1
  No | 15
Autism Mental Status Exam [Mean (Standard Deviation); unit: score on a scale] — The AMSE is an observational assessment that looks at 8 items of social, communicative and behavioral functioning in individuals with Autism Spectrum Disorder, with each item yielding a potential score of 0, 1 or 2, with range of 0-16. Higher scores indicate greater levels of impairment.
  score on a scale | 9.96 (2.29)
Presence of Co-morbid Psychiatric Disorders [Number; unit: participants]
  Autism Spectrum Disorder | 7
  BiPolar Disorder | 0
  Attention Deficit Disorder | 1
  Obsessive Compulsive Disorder | 0
  Other | 4
BSID-4 NVDQ [Mean (Standard Deviation); unit: score on a scale] — Bayley Scales of Infant Development-4 (BSID-4) is used to measure the developmental functioning of children aged 1 to 42 months.
  The Non-Verbal Developmental Quotient (NVDQ) is derived from the Cognitive scale of the BSID-4 and focuses on tasks that require no verbal responses.
  Each non-verbal task is scored and the raw scores are summed up and converted to a quotient comparing the child's developmental age to their chronological age This standardization allows comparison across children of different ages. Population: Participants who could not be assessed on the Stanford-Binet Intelligence (SB-5) due to their developmental level were assessed using the Bayley Scales of Infant Development instead.
  score on a scale
    number analyzed (Participants) | 14
    (all) | 11.602 (7.3599)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: To examine the incidence, severity and frequency of adverse events (AEs), including serious adverse events (SAEs) during treatment with NNZ-2591.
Time Frame: 13 weeks
Population: Safety population - all participants receiving at least one dose of NNZ-2591
Measure: Count of Participants; unit: Participants
Groups:
- NNZ-2591: All enrolled participants
Arm/Group | NNZ-2591
Number analyzed (Participants) | 16
Participants
  Participants with TEAE | 15
  Participants with Serious TEAE | 0
  Participants who discontinued due to TEAE | 4
  Participants with mild TEAE as highest intensity | 12
  Participants with moderate TEAE as highest intensity | 3
  Participants with severe TEAE as highest intensity | 0

2. Primary Outcome: Pharmacokinetic - Mean AUC24
Description: Approximately nine sparse pharmacokinetic (PK) samples were collected from each participant under steady-state conditions. These samples were taken at pre-dose, 1-3 hours post-dose, and/or 4-7 hours post-dose during Weeks 2, 6, and 13. The individual pharmacokinetic parameters for NNZ-2591, including half-life (t1/2) and area under the curve over 24 hours (AUC24), were derived using subject-level concentration-time profiles from the study population model.
Time Frame: Pre-dose, 1-3 h post-dose and/or 4-7 h post-dose at Weeks 2, 6 and 13.
Population: All participants enrolled in this study who receive the study drug through to the morning dose of Week 2 (Visit 5) as a minimum, and who underwent PK sample collection at least one of the specified post-dose time point(s).
Measure: Mean (Standard Deviation); unit: ug.h/mL
Groups:
- NNZ-2591: PK population:
  All participants enrolled in this study who receive the study drug through to the morning dose of Week 2 (Visit 5) as a minimum, and who undergo PK sample collection at least one of the specified post-dose time point(s).
Arm/Group | NNZ-2591
Number analyzed (Participants) | 16
ug.h/mL | 305 (56.1)

3. Primary Outcome: Pharmacokinetic - t1/2
Description: as for outcome 2
Time Frame: Pre-dose, 1-3 h post-dose and/or 4-7 h post-dose at Weeks 2, 6 and 13.
Population: All participants enrolled in this study who receive the study drug through to the morning dose of Week 2 (Visit 5) as a minimum, and who undergo PK sample collection at least one of the specified post-dose time point(s).
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NNZ-2591
Number analyzed (Participants) | 16
hours | 7.17 (1.64)

4. Secondary Outcome: Pitt Hopkins Syndrome-specific Clinical Global Impression Scale (CGI-I) - Overall Improvement
Description: Pitt Hopkins Syndrome-specific Clinical Global Impression Scale (CGI-I) - Overall Improvement. Score on a Likert scale (1-7) where lower scores are better.
Time Frame: CGI-I was assessed at weeks 6, 13/EOT & 15. Overall improvement scores relate to week 13/EOT visit.
Population: Modified intention to treat (MITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Modified Intention to Treat: All participants in the ITT population who completed treatment and completed the EOT visit.
  ITT populations consists of all participants deemed eligible and enrolled into the study.
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 2.6 (0.92)
Statistical Analysis 1: Comparison: Modified Intention to Treat; Descriptive statistics were used to summarize the data. For total scores, waterfall plots and histograms/bar charts were created at the EOT visit with plots for all participants; Test type: Other; p = .0039, Wilcoxon Signed rank; null median = 4, not 0

5. Secondary Outcome: Caregiver Impression of Improvement: Overall Score
Description: Caregiver Impression of Improvement: Overall Score. Measured on a 7 point Likert scale (1-7) where lower scores are better.
Time Frame: CIC was assessed at Week13/EOT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 3.0 (1.00)
Statistical Analysis 1: Comparison: Modified Intention to Treat; Descriptive statistics were used to summarize the data. For total scores, waterfall plots, and histograms were created at the EOT visit with plots for all participants; Test type: Other; p = 0.0234, Wilcoxon Signed rank; null median = 4, not 0

6. Secondary Outcome: Pitt Hopkins Syndrome-specific Clinical Global Impression Scale - Severity (CGI-S) - Overall Score
Description: Pitt Hopkins syndrome-specific Clinical Global Impression Scale - Severity (CGI-S) - Change from baselines on overall Score based on a 7 point Likert scale (1-7) where lower scores are better.
Time Frame: Change in score assessed from baseline (visit 3, week 0) to visit 16 (week 13/EOT).
Population: Modified intention to treat (MITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | -0.5 (0.52)
Statistical Analysis 1: Comparison: Modified Intention to Treat; Efficacy endpoints were analyzed using a Wilcoxon signed rank test on the paired participant data from baseline to EOT (Visit 16), when applicable. Baseline values were based on the average non-missing values of visits 1, 2, and 3 for assessments collected at more than one visit during the Screening/Baseline period; Test type: Other — Change from baseline; p = 0.0313, Wilcoxon Signed rank

7. Secondary Outcome: Caregiver Top 3 Concerns
Description: Caregiver Top 3 Concerns: Change from baseline in Average Concern Severity. The average concern severity defined as the average of the severity scores for the three concerns evaluated at a given visit, and was calculated as long as at least one concern was useable for analysis at the visit. Scores range from 0 - 10 with higher scores indicating greater concern severity. A negative change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in average concern severity.
Population: Modified intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | -1.606 (1.5385)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.0039, Wilcoxon Signed rank

8. Secondary Outcome: MacArthur-Bates Communicative Development Inventory (MB-CDI)
Description: MacArthur-Bates Communicative Development Inventory (MB-CDI): Words Understood Domain. Scores ranges from 0-396, with higher scores indicating greater language ability. A positive change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 15.9 (42.07)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — change from baseline; p = 0.1934, Wilcoxon Signed rank

9. Secondary Outcome: Observer-Reported Communication Ability (ORCA)
Description: Observer-Reported Communication Ability (ORCA): Change from baseline in Modified t-score. The ORCA measures an individual's communication abilities based on observations made by caregivers, parents, or other relevant observers, and is based on 4 domains: Expressive Communication, Receptive Communication, Social Communication, and Pragmatic Language Skills.
  Scores range from 25.8 - 83.8, with higher scores indicating greater communication ability. A positive change from baseline indicates improvement. A T-score standardizes the individual's performance relative to a normative sample. It typically has a mean of 50 and a standard deviation of 10.
  T score = 50 + 10 × (X-µ)/σ Where: X is the individual's raw score μ is the population mean σ is the standard deviation
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in Total Score.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
T-score | 1.97 (8.963)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.7480, Wilcoxon Signed rank

10. Secondary Outcome: Aberrant Behavior Checklist-2 (ABC-2)
Description: Aberrant Behavior Checklist-2 (ABC-2): Change from baseline in Total Score. Range of scores is 0-174, with higher scores indicating more behavioral issues. A negative change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in total score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | -4.8 (14.15)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.3203, Wilcoxon Signed rank

11. Secondary Outcome: CSHQ
Description: Child Sleep Habits Questionnaire (CSHQ). Total Score. Change from baseline. Range of scores was (33-99) with higher scores being worse.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in total score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 0.4 (1.79)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — change from baseline; p = 0.3574, Wilcoxon Signed rank

12. Secondary Outcome: GIHQ
Description: Gastrointestinal Health Questionnaire (GIHQ). Change from baseline in total frequency score. Range of scores was (0-197) with higher scores being worse.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in total frequency score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | -6.3 (21.83)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.4131, Wilcoxon Signed rank

13. Secondary Outcome: Vineland Adaptive Behavior Scales-3, Interview Version
Description: Vineland Adaptive Behavior Scales-3 (VABS-3), Interview version, Change from baseline in Adaptive Behavior Composite Standard Score. Scores range from 20 - 140 with higher scores indicating greater functional abilities. A positive change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in composite standard score.
Population: one participant completed baseline VABS-3 but did not complete VABS-3 at EOT visit. Hence number analysed is only 10.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 10
score on a scale | 0.0 (2.36)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — change from baseline; p = 0.9063, Wilcoxon Signed rank

14. Secondary Outcome: Modified Two-minute Walk Test
Description: Modified two-minute walk test. Change from baseline in distance travelled (m) on 2 minute walk test. The test was only administered for participants who were ambulatory and able to complete the assessment. A positive score on change from baseline indicates improvement in distance walked.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in distance travelled on two minute walk test.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 8
meters | 8.704 (25.7178)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 1.00, Wilcoxon Signed rank

15. Secondary Outcome: QI-Disability
Description: Quality of Life Inventory-Disability (QI-Disability). Overall Score change from baseline. Scores range from 0 - 100 with higher scores indicating better quality of life. A positive change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in overall score score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | -1.672 (9.8493)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.7002, Wilcoxon Signed rank

16. Secondary Outcome: ICND
Description: Impact of Childhood Neurological Disability (ICND)-Overall quality of life rating, change from baseline. Score ranges from 1 - 6, with a higher score indicating better quality of life. A positive change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in overall quality of life rating score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 0.5 (1.44)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other — Change from baseline; p = 0.3750, Wilcoxon Signed rank

17. Secondary Outcome: Behavior Problems Inventory - Short Form
Description: Change from baseline in Behavior Problems Inventory - Short Form Total Frequency Score. Scores range from 0-120, with higher scores indicating greater frequency in behavior problems. A negative change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in Total Frequency score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 3.2 (15.45)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.7695, Wilcoxon Signed rank

18. Secondary Outcome: Bayley Scales of Infant Development (BSID-4): Non Verbal Development Quotient (NVDQ)
Description: Change from baseline in Non Verbal Development Quotient (NVDQ). Scores range from 40 - 160, with higher scores indicating greater development. A positive change from baseline indicates improvement.
Time Frame: Change from baseline (visit 3, week 0) to visit 16/EOT (week 13) in NVDQ score.
Population: Standard domain scores only calculated for participants 42 months of age and younger.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Modified Intention to Treat
Number analyzed (Participants) | 11
score on a scale | 0.444 (2.4685)
Statistical Analysis 1: Comparison: Modified Intention to Treat; [analysis description as in outcome 6, analysis 1]; Test type: Other; p = 0.2402, Wilcoxon Signed rank

ADVERSE EVENTS:
Time Frame: 15 weeks for each participant starting on the day of first dosing
Groups:
- NNZ-2591: All enrolled participants who received at least one dose of IMP
Arm/Group | NNZ-2591
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNZ-2591 (N=16)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Somnolence (Nervous system disorders) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Gastroenteritis - viral (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Covid-10 (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Breath Odour (Gastrointestinal disorders) | 1 (1)
Faeces Hard (Gastrointestinal disorders) | 1 (1)
Tongue Dry (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Intentional Self Injury (Psychiatric disorders) | 1 (1)
Middle Insomnia (Psychiatric disorders) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Refraction Disorder (Eye disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05025332/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05025332/SAP_003.pdf